CLINICAL TRIAL: NCT01455506
Title: PRO#0118: A Phase I Study of Decitabin in Combination With Fludarabin and Busulfan as a Reduced Intensity Conditioning Regimen for the Treatment of Myeloid Malignancies
Brief Title: PRO#0118: Decitabine Plus Mini Flu-Bu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Decitabine plus mini-FluBu
Record Dates: First submitted 2011-06-02; First posted 2011-10-20 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Bone Marrow Transplant; Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine; fludarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine with fludarabine and busulfan (Experimental): decitabine with fludarabine and busulfan in the setting of allogeneic stem cell transplantation
  Interventions: Drug: Decitabine plus Fludarabine and Busulfan

INTERVENTIONS:
Drug: Decitabine plus Fludarabine and Busulfan — * Decitabine will be administered at a dose of 60 mg/m2 IV daily based on adjusted body weight for patient >20% above ideal body weight
  * Fludarabine will be administered at a dose of 30/mg/m2 IV daily for 5 days starting on transplant day -7.
  * Busulfan will be administered at a dose of 130 mg/m2 IV daily for 2 days on transplant days -4 and -3.
  Patients will also receive rabbit antithymocyte globulin (Thymoglobulin) at a dose of 2 mg/kg IV daily for 3 days on transplant days -4, -3, and -2.
  Hematopoietic cells will be infused on day 0.

SUMMARY:
This is a single institution study of combining decitabine with fludarabine and busulfan in the setting of allogeneic stem cell transplantation. A study population of 20 subjects will be enrolled from The John Theurer Cancer Center at Hackensack University Medical Center. Subjects who are eligible to receive allogeneic hematopoietic stem cell transplantation according to the eligibility criteria will be consented and enrolled. Subjects will receive treatment with decitabine followed by reduced intensity fludarabine and busulfan prior to allogeneic stem cell transplantation. Subjects will be followed until 1 year post transplantation to assess stability of engraftment, toxicity, progression free survival, and disease response

DETAILED DESCRIPTION:
Aberrant DNA methylation patterns are commonly found in malignant cells. Hypermethylation of gene promotes sequences in cancer cells resulting in transcriptional silencing of tumor suppressor genes and contributing to malignant transformation. Hypomethylating agents have been explored for the treatment of cancers such as acute myelogenous leukemia and myelodysplastic syndrome. In vitro inhibition of methylation using azanucleosides results in differentiation of transformed myeloid cells. In vivo these agents induce DNA methylation of malignant myeloid cells. The most potent DNA methylating agent currently available, decitabine, is effective in patients with myelodysplastic syndrome (MDS) and acute myelogenous leukemia (AML). About 30% of patients with MDS and an abnormal karyotype will have normalization of their karyotype after receiving the drug.

The myelodysplastic syndromes are a heterogeneous group of clonal hematologic disorders characterized by bone marrow failure and proliferation of myeloblastic leukemia cells. Patients with MDS develop cytopenias as a result of ineffective hematopoiesis. These cytopenias are believed to be a result of an increase in apoptosis resulting in an increase in futile cell cycling. In addition, the apparently mature and differentiated hematopoietic cells in patients with MDS are functionally impaired. Granulocytes have decreased myeloperoxidase activity and platelets have impaired function. Therapy for MDS includes supportive care geared mostly to transfusional support. Allogeneic transplantation has been shown to offer the possibility of long-term remission and remains the only curative option for patients with MDS. The development of reduced intensity conditioning regimens expanded the scope of allogeneic transplantation for older patients with MDS. A very large retrospective analysis by the European Blood and Marrow Transplantation Group compared the outcome of 836 patients with MDS treated with either a reduced-intensity conditioning regimen or a conventional regimen before allogeneic transplantation. The 3-year probabilities of progression-free and overall survival were similar in both groups, with a 3-year relapse rate being significantly higher in the reduced-conditioning group, offset by a significantly reduced probability of non-relapse mortality. This demonstrates the importance of the preparative regimen in preventing relapse in this setting.

Acute myeloid leukemia accounts for over 9,000 deaths yearly in the United States. The WHO classification of AML incorporates and interrelated morphology, cytogenetics, molecular genetics and immunologic markers in an attempt to construct a classification that is clinically and prognostically valid. Under this classification the requisite blast percentage in the marrow is > 20%. Hematopoietic stem cell transplantation is an established therapeutic modality in patients with AML. An alloreactive immunotherapeutic effect of donor cells has been demonstrated.

No other established therapy applied during complete remission offers as strong an anti-leukemic effect. Transplant-related morbidity and mortality, however, remain obstacles in the successful application of this treatment. More recently, reduced-intensity conditioning has been applied as a therapy for AML. Reduced-intensity conditioning, which includes potent immunosuppressive agents in addition to anti-leukemic agents, effectively permits engraftment of donor hematopoietic stem cells. Several studies have demonstrated that the morbidity and mortality are less with these regimens compared to myeloablative conditioning. While the reduced intensity of the conditioning regimen has resulted in reduced non-relapse mortality in patients with AML, some studies have suggested a concomitant increase in relapse as a consequence of lowering the intensity of the cytotoxic agents. New conditioning regimen that may increase the anti-leukemic effect while maintaining the reduced-intensity regimen toxicity profile are therefore, needed.

Decitabine is a deoxycytidine analog that rapidly enters into cells by a nucleoside-specific transport mechanism. It is then phosphorylated by deoxycytidine kinase and converted to the active triphosphate form, 5AZA-dCTP, a substrate for DNA polymerase alpha. 5AZA-dCTP is incorporated into DNA and inhibits DNA methylation as inactivating DNA methyltransferase. Decitabine is s-phase specific. A recent study randomized 170 patients with MDS to receive either decitabine or best supportive care. Patients who were treated with decitabine achieved a significantly higher overall response rate (17%) including complete responses (9%), compared with supportive care (0%). Responses were durable and were associated with transfusion independence. Patients treated with decitabine had a trend toward a longer median time to acute myelogenous leukemia (AML) progression or death compared with patients who received supportive care alone. Responses in AML have also been demonstrated with 14% complete responses and 8% partial responses in one study . Decitabine has been used in combination with cyclophosphamide and busulfan as preparative regimen in patients with AML. This regimen was associated with a high response rate, with 40% of patients with AML being still in remission more than three years after transplantation. The total dose of decitabine ranged from 400 mg/m2 to 800 mg/m2. No decitabine dose-limiting toxicity was documented. The combination of fludarabine and busulfan has been well established as a transplant regimen and is associated with a reduced regimen-related toxicity. The combination of fludarabine and busulfan is the current standard of care for AML patients undergoing allogeneic transplantation at HUMC. In this study the investigators will be using the combination of reduced-intensity fludarabine and busulfan along with decitabine 300 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myelogenous leukemia or myelodysplastic syndrome being considered for transplantation.
* Age 45 to 80 years or < 45 with co-morbidity including: disease not in remission
* No uncontrolled infections.
* Patients shall have a 6/6 HLA-compatible related donor or an 8/8 -HLA-compatible unrelated donor.
* KPS 70-100%
* Creatinine < 1.6 X ULN (unless age < 45 yrs)
* Serum Bilirubin < 2.5 X ULN
* Capable of giving informed consent and have signed the informed consent form.
* Cardiac EF > 50% or cardiac clearance
* Pulmonary DLCO > 50% or pulmonary clearance

Exclusion Criteria:

* Untreated CNS leukemia
* Active hepatitis or other untreated infections

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of decitabine in combination with fludarabine and busulfan prior to allogeneic stem cell transplantation on the rate of primary graft rejection | up to 1 year post transplantation
  Graft failure defined by the presence of <10% donor lymphoid cells on peripheral blood analysis performed on post transplant day 84(+/- 10 days) in patients who have not relapsed will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, MD, Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center
Locations (1):
- Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey, United States